CLINICAL TRIAL: NCT00528073
Title: A Phase II, Multicentre, Double-blind, Randomised, Dose Range Finding Placebo Controlled Study of Rifaximin-EIR Tablet: Clinical Effectiveness and Tolerability in the Treatment of Moderate, Active Crohn's Disease
Brief Title: Placebo Controlled Study of 3 Doses of Rifaximin-EIR Tablet to Treat Moderate, Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Dr Pier Alessandro Monici Preti MD, Alfa Wassermann S.p.A.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RETIC/03/06; EudraCT: 2007-001014-17
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Crohn's Disease
Keywords: Rifaximin-EIR; Crohn's disease; remission
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): Rifaximin-EIR tablet 1x400 mg + Placebo 2 tablets bid
  Interventions: Drug: Rifaximin-EIR
- B (Experimental): Rifaximin-EIR tablet 2x400 mg + Placebo 1 tablet bid
  Interventions: Drug: Rifaximin-EIR
- C (Experimental): Rifaximin-EIR tablet 3x400 mg bid
  Interventions: Drug: Rifaximin-EIR
- D (Placebo Comparator): Placebo 3 tablets bid
  Interventions: Drug: Rifaximin-EIR

INTERVENTIONS:
Drug: Rifaximin-EIR — Comparison of 800 mg, 1600 mg and 2400 mg Rifaximin-EIR versus placebo in the treatment of active moderate Crohn's disease
  Other Names: GRACE

SUMMARY:
This study aims to determine which of 3 doses of a non-absorbable antibiotic Rifaximin is most effective in treating active moderate Crohn's disease. Rifaximin tablets are already marketed in some European countries and the USA to treat traveller's diarrhoea. A new gastro-resistant form of Rifaximin called Rifaximin-Extended Intestinal Release (EIR) will be used in this study. These tablets dissolve in the stomach,releasing gastro-resistant granules which pass into the intestines and deliver Rifaximin directly to the site of the disease. Rifaximin is not absorbed, making it more effective and greatly reducing the frequency of side effects.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Crohn's disease localised in the ileum and/or colon, documented either radiologically or endoscopically at least 3 months previously;
* patients with a CDAI of ≥ 220 to ≤ 400;
* patients capable of and willing to conform to the study protocol;
* patients who have provided signed and dated written informed consent.

Exclusion Criteria:

* patients potentially needing immediate surgery for Crohn's disease, including patients with occlusive symptoms and/or stenotic tract with dilation above;
* patients with active perianal Crohn's disease;
* patients with other infectious, ischemic, or immunological diseases with gastrointestinal involvement;
* patients with symptoms attributed to Short Bowel Syndrome or previous surgery;
* patients with stoma;
* patients affected by upper gastro-intestinal disease (gastro-duodenum-jejunum Crohn's disease) alone or in combination with colitis or ileitis;
* patients treated with: oral steroids and budesonide less than 30 days prior to screening; i.v. steroids less than 30 days prior to screening; antibiotics (such as metronidazole, tinidazole, ciprofloxacin, clarithromycin) less than 15 days prior to screening;
* rectal steroids less than 30 days prior to the screening visit;
* anti-tumour necrosis factor (anti-TNF) and other biological therapies less than 6 months prior to the screening visit;
* pregnant women or nursing mothers;
* females of childbearing age (unless surgically sterile) without a negative urine pregnancy test at screening and at enrolment;
* patients with severe hepatic insufficiency (Child C);
* patients with severe cardiac insufficiency (NYHA - New York Heart Association classes 3 - 4);
* patients with known hypersensitivity to Rifaximin;
* any condition or circumstance that would prevent completion of the study or interfere with analysis of study results, including a history of drug or alcohol abuse, mental illness or non-compliance with treatments or visits, with immunological (including HIV infection), haematological or neoplastic disease;
* withdrawal of informed consent;
* patients who have used any investigational drug (except biological therapies) within 3 months prior to screening;
* patients who have donated 250 ml or more of blood in the last 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Clinical remission (Crohn's Disease Activity Index < 150 points) | After 12 weeks of treatment

SECONDARY OUTCOMES:
Clinical response (reduction of baseline CDAI score by 100 points or more) | Any time during the 12 weeks of treament
Clinical response (reduction of baseline CDAI by 70 points or more) | At any time during the 12 weeks of treatment
Time to obtain clinical response and remission | During the 12 weeks of treatment
Maintenance of clinical remission | 2 weeks after the end of the 12 weeks of treatment
Maintenance of clinical remission | 12 weeks after the end of the 12 weeks of treatment
Number of treatment failures | During the 12 weeks of treatment
Definition of therapeutic dose to be used in subsequent phase III trials. | After statistical analysis of the results
Adverse events | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Pier Alessandro Monici Preti, MD, Study Chair — Alfa Wassermann; Maria Grimaldi, MD, Study Director — Alfa Wassermann; Cosimo Prantera, MD, Principal Investigator — S. Camillo - Forlanini Hospital
Locations (57):
- France (5):
  - CHU Amiens, Hôpital Nord, Amiens
  - Hôpital Saint André, Bordeaux
  - CHU Grenoble, Hôpital Michallon, Grenoble
  - CHU de Nice, Hôpital de l'Archet II, Nice
  - CHU de Rouen, Hôpital Charles Nicolle, Rouen
- Germany (8):
  - Charité Campus Mitte, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Interdisziplinäres Facharztzentrum, Zentrum für Viszerale- und Ernährungsmedizin, Frankfurt am Main
  - Medizinische Hochschule Hannover, Hanover
  - Abteilung Gastroenterologie, Charité Campus Benjamin Franklin, Hindenburgdamm 30, Berlin
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsklinikum Mannheim, Mannheim
  - Gastroenterological Group Practice, Minden
- Hungary (6):
  - Allami Egeszsegugyi Kozpont, MAV-Rendeszeti Szervek-Honvedseg Egyesitett Korhaza, Budapest
  - Debreceni Egyetem Orvos és Egészégtudományi Centrum II. Belgyógyászati Klinika, Debrecen
  - Békés Megyei Kèpviselőtestület, Pándy Kálmán Kórház, III. Belgyógyászat, Gyula
  - Szegedi Tudományegyetem, Általános Orvostudományi Kar, I. sz. Belgyógyászati Klinika, Szeged
  - Tolna Megyei Önkormányzat Balassa János Kórhaz, II. Belgyógyászat, Szekszárd
  - Jávorszky Ödön Kórház, Gasztroenterológiai Osztály, Vác
- Israel (5):
  - Bnai Zion Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (10):
  - Casa Sollievo della Sofferenza IRCCS, San Giovanni Rotondo, Foggia
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Azienda Ospedaliera-Universitaria di Bologna - Policlinico S. Orsola-Malpighi, Bologna
  - A.O. Luigio Sacco U.O gastraneterologia, via G.B. grassi 74, Milan
  - Azienda Ospedaliera Padova, Padua
  - Azienda Ospedaliera Universitaria Policlinico di Torvergata, Rome
  - Azienda Ospedaliera "San Camillo-Forlanini", Rome
  - Policlinico "A,. Gemelli", Rome
  - Azienda Ospedaliera S. Giovanni Battista Molinette, Turin
  - Ospedale Mauriziano "Umberto I", Turin
- Poland (8):
  - 10 Wojskowy Szpital Kliniczny z Polikliniką, Bydgoszcz
  - Wojewódzki Szpital Specjalistyczny im. Najświętszej Maryi Panny, Częstochowa
  - Szpital Specjalistyczny Św. Wojciecha- Adalberta, Gdansk
  - Samodzielny Publiczny Centralny Szpital Kliniczny Im Prof. Kornela Gibinskiego Ślaskiej Akademii Medycznej, Katowice
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnętrznych i Administracji, Warsaw
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie, Warsaw
  - Akademicki Szpital Kliniczny Im. Jana Mikulicza-Radeckiego, Wroclaw
- Russia (15):
  - Russian Center of Functional Surgical Gastroenterology, Krasnodar
  - Sechenov Moscow Medical Academy, Moscow
  - State Scientific Centre of Coloproctology, Moscow
  - City Clinical Hospital # 24, Moscow
  - Moscow Regional Research Clinical Institute n.a. M.F. Vladimirsky, Moscow
  - Nizhny Novgorod Regional Clinical Hospital, Nizhny Novgorod
  - Novosibirsk State Medical University City Hospital #7, Novosibirsk
  - Rostov State Medical University City Hospital # 20, Rostov-on-Don
  - City Polyclinic # 38, Saint Petersburg
  - Military Medical Academy, Saint Petersburg
  - Sokolov Clinical Hospital #122, Saint Petersburg
  - St. Petersburg Mechnikov State Medical Academy, Saint Petersburg
  - MAPO, City Hospital # 26, Saint Petersburg
  - St. Petersburg MAPO, City Hospital #31, Saint Petersburg
  - Yaroslavl Regional Clinical Hospital, Yaroslavl

REFERENCES:
- [Background] Prantera C, Lochs H, Campieri M, Scribano ML, Sturniolo GC, Castiglione F, Cottone M. Antibiotic treatment of Crohn's disease: results of a multicentre, double blind, randomized, placebo-controlled trial with rifaximin. Aliment Pharmacol Ther. 2006 Apr 15;23(8):1117-25. doi: 10.1111/j.1365-2036.2006.02879.x. PMID 16611272
- [Derived] Prantera C, Lochs H, Grimaldi M, Danese S, Scribano ML, Gionchetti P; Retic Study Group (Rifaximin-Eir Treatment in Crohn's Disease). Rifaximin-extended intestinal release induces remission in patients with moderately active Crohn's disease. Gastroenterology. 2012 Mar;142(3):473-481.e4. doi: 10.1053/j.gastro.2011.11.032. Epub 2011 Dec 6. PMID 22155172